CLINICAL TRIAL: NCT01651520
Title: Prognosis Value of the Neuronal Damage Detected by Positrons Emission Tomography (PET) With 11C-Flumazenil in Early Multiple Sclerosis.
Brief Title: Prognosis Value of the Neuronal Damage in Early Multiple Sclerosis
Acronym: Flumatep_2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IDRCB 2011-A00836-35; P100126 (Other: APHP)
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
Keywords: Neurodegeneration; Disability; Cognition; Prognosis
MeSH Terms: conditions — Multiple Sclerosis; Nerve Degeneration | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Relapsing patients < 5 years (Experimental): Relapsing patients < 5 years
  Interventions: Drug: PET with 11C-Flumazenil
- relapsing patients < 10 years (Experimental): relapsing patients < 10 years
  Interventions: Drug: PET with 11C-Flumazenil
- primary progressive patients < 10 years (Experimental): primary progressive patients < 10 years
  Interventions: Drug: PET with 11C-Flumazenil
- healthy volunteers (Other): healthy volunteers
  Interventions: Drug: PET with 11C-Flumazenil

INTERVENTIONS:
Drug: PET with 11C-Flumazenil — PET with 11C-Flumazenil.

SUMMARY:
In this study the investigators will use PET and 11C-Flumazenil to visualize and quantify neuronal injury in the cortex and the deep gray matter of Multiple Sclerosis patients at an early stage. The investigators will follow up patients to determine the prognostic value of this neuronal injury.

DETAILED DESCRIPTION:
It is now well admitted that multiple sclerosis (MS), which is an inflammatory demyelinating disease of the central nervous system (CNS) is not restricted to white matter, but also involves grey matter, either the cortex or the deep grey matter. The progression of grey matter atrophy measured by MRI during disease course represents an interesting prognosis marker for long term progression, but this marker lack sensitivity and is hard to interpret at the individual level.

In the EAE animal models, an early neuronal damage has been described, characterized both by a synaptic and dendritic loss and by a neuronal apoptosis.

These data strongly suggest that the occurrence of an early neuronal damage during MS course could represent a major prognosis marker. Therefore there is a crucial need for the development of imaging techniques, aimed at visualizing and quantifying neuronal damage in early MS. To date MRI techniques are not able to specifically assess neuronal pathology in vivo.

In this prospective project we will determine the chronology of appearance and the prognosis value of the neuronal damage measured by PET with 11C-Flumazenil, concerning further grey matter atrophy progression and disability progression among a cohort of MS patients with recent onset.

Four groups of subjects will be included: i) patients with a RRMS evolving since less than 5 years (revised Mc Donald criteria, n=20); ii) patients with a RRMS evolving since more than 5 years and less than 10 years (n=20); iii) patients with a primary progressive MS (PPMS) evolving since less than 10 years (n=20); iv) Healthy volunteers matched for age and sex (2/3 matched with RRMS patients; 1/3 matched with PPMS patients).

Each subject will pass a neurologic examination, a neuropsychological testing, a first PET examination with 11C-Flumazenil, a multimodal MRI, with conventional sequences (3DT1, 3D T2 and FLAIR, pre and post contrast T1) and non conventional sequences (MTR, DTI, protonic spectroscopy).

All patients will be followed prospectively with one visit/year consisting in clinical neurological, and neuropsychological evaluations as well as multimodal MRI.

For healthy volunteers a second PET 11C-Flumazenil will also be performed to assess reproducibility and evolution (50% after 1 month, 50% after 1 year).

This study will allow to assess on a larger sample followed prospectively (5 years) the prognosis value of abnormalities detected and quantified by PET with 11C-Flumazenil on further grey matter atrophy progression on MRI and disability progression (EDSS, MSFC, cognitive status). It will also precise the chronology of appearance and the evolution of neuronal damage in MS, and determine the reproducibility of this technique. Results should provide a new and more efficient prognosis marker for early MS.

ELIGIBILITY:
Inclusion Criteria:

Four groups of subjects will be included:

* patients with a RRMS evolving since less than 5 years (revised Mc Donald criteria, n=20);
* patients with a RRMS evolving since more than 5 years and less than 10 years (n=20);
* patients with a primary progressive MS (PPMS) evolving since less than 10 years (n=20);
* Healthy volunteers matched for age and sex (2/3 matched with RRMS patients; 1/3 matched with PPMS patients).

Exclusion Criteria:

* Lack of social insurance
* Pregnancy
* Age > 55
* Therapy with benzodiazepine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
neuronal imaging | 2 years
  Prognosis value of the neuronal imaging on 2 years evolution (atrophy and EDSS)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Stankoff, MD, PhD, Principal Investigator — APHP
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

REFERENCES:
- [Derived] Ricigliano VAG, Louapre C, Poirion E, Colombi A, Yazdan Panah A, Lazzarotto A, Morena E, Martin E, Bottlaender M, Bodini B, Seilhean D, Stankoff B. Imaging Characteristics of Choroid Plexuses in Presymptomatic Multiple Sclerosis: A Retrospective Study. Neurol Neuroimmunol Neuroinflamm. 2022 Oct 13;9(6):e200026. doi: 10.1212/NXI.0000000000200026. Print 2022 Nov. PMID 36229188